CLINICAL TRIAL: NCT01070472
Title: Efficacy and Safety of Titrated Oral Misoprostol Solution for Labor Induction at Term
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. debbie Robinson, Dr, University of Manitoba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2009:149
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Labor Induction at Term
Keywords: labor induction at term using a titrated oral misoprostol solution
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Misoprostol — titrated oral misoprostol solution

SUMMARY:
The purpose of this study is to determine whether a titrated solution of oral Misoprostol is safe and effective at inducing labor at term, regardless of Bishop Score.

ELIGIBILITY:
Inclusion Criteria:

1. term,
2. singleton
3. no contraindication to prostaglandins
4. vertex
5. no exposure to vaginal prostaglandins in the index pregnancy

Exclusion Criteria:

1. parity > 3
2. severe PIH: BP> 160/100, abnormal LFT's, proteinuria >1g/day
3. previous uterine surgery
4. regular uterine contractions
5. maternal age > 45
6. twins

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of vaginal delivery within 24 hours | 24 hours

SECONDARY OUTCOMES:
Uterine hyperstimulation rate | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: debbie J Robinson, MD FRCSC, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada